CLINICAL TRIAL: NCT06468930
Title: Efficacy of Adjunctive Low-Level Light Therapy to Intense Pulsed Light for Meibomian Gland Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0666/66
Record Dates: First submitted 2024-03-28; First posted 2024-06-21 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-02

CONDITIONS: MGD-Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Low-Level Light Therapy; Intense Pulsed Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ALLLT + IPL group (Experimental): Participants will receive a session of IPL therapy followed by LLLT therapy, once weekly for 4 weeks (total 4 treatment sessions). The IPL therapy will be performed using the Eye-light® with Optimal Power Energy® (Espansione Marketing S.p.A., Bologna, Italy), which emits the light at a wavelength of 600 nm IPL system with fluence ranging from 10 to 16 J/cm2 per eye depending on the Fitzpatrick skin scale. During IPL treatment 5 flashes of light will be applied to the skin around the eye using a handheld device; 3 along the inferior orbital rim, 1 at the lateral canthus, and 1 applied horizontally along the inferior orbital rim. The LLLT therapy will be delivered using the Light Modulation® special facial mask (Espansione Marketing S.p.A., Bologna, Italy) which will be placed on the participant's face for 15 minutes. The mask has the shape of a half-face and will emit a red light in a light-emitting diode (LED) system.
  Interventions: Device: Low-level light therapy (LLLT); Device: Intense pulsed light (IPL)
- IPL alone group (Active Comparator): The IPL alone group will receive only a session of IPL therapy, once weekly for 4 weeks (total 4 treatment sessions). The IPL therapy will be performed using the Eye-light® with Optimal Power Energy® (Espansione Marketing S.p.A., Bologna, Italy), which emits the light at a wavelength of 600 nm IPL system with fluence ranging from 10 to 16 J/cm2 per eye depending on the Fitzpatrick skin scale. During IPL treatment 5 flashes of light will be applied to the skin around the eye using a handheld device; 3 along the inferior orbital rim, 1 at the lateral canthus, and 1 applied horizontally along the inferior orbital rim, similar to the combined group. Additionally, the special facial mask will also be placed on the participant's face for 15 minutes with no light power applied.
  Interventions: Device: Intense pulsed light (IPL)

INTERVENTIONS:
Device: Low-level light therapy (LLLT) — LLLT therapy will be delivered using the Light Modulation® special facial mask (Espansione Marketing S.p.A., Bologna, Italy) which will be placed on the participant's face for 15 minutes. The mask has the shape of a half-face and will emit a red light in an LED system. The device has an emission power of 100 The mask has the shape of a half-face and will emit a red light in a light-emitting diode (LED) system. The device has an emission power of 100 milliwatts per square centimeter.
  Arms: ALLLT + IPL group
Device: Intense pulsed light (IPL) — The IPL therapy will be performed using the Eye-light® with Optimal Power Energy® (Espansione Marketing S.p.A., Bologna, Italy), which emits the light at a wavelength of 600 nm IPL system with fluence ranging from 10 to 16 J/cm2 per eye depending on the Fitzpatrick skin scale. During IPL treatment 5 flashes of light will be applied to the skin around the eye using a handheld device; 3 along the inferior orbital rim, 1 at the lateral canthus, and 1 applied horizontally along the inferior orbital rim

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of adjunctive low-level light therapy (LLLT) to intense pulsed light (IPL) versus intense pulsed light (IPL) alone for the treatment of meibomian gland dysfunction (MGD).

The main question it aims to answer is does the adjunctive of low-level light therapy (LLLT) to intense pulsed light (IPL) provide more beneficial treatment effects than intense pulsed light (IPL) alone in treating meibomian gland dysfunction (MGD) patients?

Participants will be randomized into 2 groups: adjunctive low-level light therapy (LLLT) to intense pulsed light (IPL) group (ALLLT +IPL) and IPL alone group.

DETAILED DESCRIPTION:
In both the IPL group and the ALLLT+IPL group, the doctor will administer IPL therapy to each participant and apply the Light Modulation® special facial mask to their faces. The assistant nurse will activate the light power, ensuring that the doctor remains blind to treatment allocation. Participants in both groups will receive a conventional treatment for MGD including warm compression and lid hygiene. Moreover, all participants will be advised to use preservative-free artificial tears 4 times daily throughout the study.

ELIGIBILITY:
Inclusion criteria:

* MGD severity level 2 and above according to the international workshop on MGD
* Fitzpatrick skin type of 1-4 according to sun sensitivity characteristics and appearance of the skin color

Exclusion Criteria:

* History of previous ocular trauma or surgery within the past six months
* Contact lens-wearing patients
* Patients with skin-pigmented lesions in the treatment area
* Pregnancy or breastfeeding patients
* Patients with any uncontrolled ocular or systemic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Lipid layer thickness (LLT) | baseline, 2 weeks, 4 weeks, 12 weeks, and 24 weeks post treatment
  Lipid layer thickness will be evaluated using Lipiview® II interferometer (TearScience®, Johnson & Johnson Vision, California, USA). The thickness of the lipid layer is then calculated from the interference pattern and expressed in interferometric color units (ICU), where 1 ICU reflects approximately 1 nm of lipid layer thickness.

SECONDARY OUTCOMES:
Meibum quality score | baseline, 2 weeks, 4 weeks, 12 weeks, and 24 weeks post treatment
  Meibum quality grade will be evaluated on central 8 glands at the lower lid with grade 0 indicating clear meibum, 1 indicating cloudy meibum, 2 indicating cloudy particulate meibum, and 3 indicating inspissated, like toothpaste meibum.
Meibum expressibility score | baseline, 2 weeks, 4 weeks, 12 weeks, and 24 weeks post treatment
  Meibum expressibility score will be evaluated on central 8 glands at the lower lid with 0 indicating all glands expressible, 1 indicating 3-4 glands expressible, 2 indicating 1-2 glands expressible, and 3 indicating no gland expressible.
Meiboscore | baseline, 2 weeks, 4 weeks, 12 weeks, and 24 weeks post treatment
  Meibography will be evaluated using Lipiview® II interferometer (TearScience®, Johnson & Johnson Vision, California, USA) Meiboscore will be graded according to meibomian gland dropout; grade 0 indicates no loss of meibomian gland, grade 1 indicates less than 25% gland loss, grade 2 indicates 25-50% gland loss, grade 3 indicates 50-75% gland loss, and grade 4 indicates more than 75% gland loss.
Tear film break-up time (TBUT) | baseline, 2 weeks, 4 weeks, 12 weeks, and 24 weeks post treatment
  TBUT will be measured using the standard fluorescein staining method.
Conjunctival and corneal staining: | baseline, 2 weeks, 4 weeks, 12 weeks, and 24 weeks post treatment
  Conjunctival and corneal staining will be evaluated using National Eye Institute (NEI) industry scale ranging from 0-33.
Ocular surface disease index (OSDI) scores | baseline, 2 weeks, 4 weeks, 12 weeks, and 24 weeks post treatment
  OSDI scores will be evaluated using a validated questionnaire, with a total score ranging from 0-100. Higher values indicating greater symptom severity; normal (<12), mild (13-22) moderate (23-32) or severe (33-100).
Tear cytokines levels | baseline and 12 weeks post treatment
  Tear samples were collected using a Schirmer strip placed at the inferior fornix without anesthesia waiting for 5 minutes, then the strip will be kept in a 2 ml centrifuge tube. The samples were stored at -20°C for further assays.

CONTACTS AND LOCATIONS:
Overall Officials: Chatchada Kharuhayothin, Principal Investigator — Ophthalmology department, Faculty of medicine, Chulalongkorn university
Locations (1):
- King Chulalongkorn memorial hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No